CLINICAL TRIAL: NCT01786044
Title: The Impact of a "Serious Game" on Improving Patient's Medication Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William Lester, Assistant in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MGH 2012-P-002093/1; PCHI MGH 2012-P-002093/1 (Other Grant/Funding Number: PCHI System Improvement Grant program)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2014-03

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: patient education; primary health care
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MasterMed (Experimental): MasterMed, an online interactive educational program
  Interventions: Behavioral: MasterMed
- Usual care (Placebo Comparator): Access to an online patient portal
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: MasterMed — An online interactive educational program
  Arms: MasterMed
Behavioral: Usual Care
  Arms: Usual care

SUMMARY:
The purpose of this study is to assess the effects of an interactive educational program delivered through a patient portal on patients' medication knowledge and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. MGH Internal Medical Associates patients
2. are age of 18 or older,
3. have at least two medications on their medication list that match our pre-selected medications,
4. have at least three medical conditions on their problem list that match our pre-selected medical conditions,
5. have at least three medications documented on their medication list, and
6. list English as their primary language.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
medication knowledge | 3 months
medication adherence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William Lester, MD, MS, Principal Investigator — Massachusetts General Hospital, Laboratory of Computer Science
Locations (1):
- Massachusetts General Hospital, Internal Medicine Associates, Boston, Massachusetts, United States